CLINICAL TRIAL: NCT00687479
Title: Clinically Useful Methods for Assessment of Insulin Sensitivity and Beta Cell Function in Women at High Risk for Gestational Diabetes: Does Race Matter?
Brief Title: Insulin Action During Pregnancy in Woman at High Risk for Gestational Diabetes
Acronym: DRM
Status: Completed | Type: Observational
Sponsor: Woman's (Other)
Collaborators: Baton Rouge Area Foundation (Other)
Responsible Party: Principal Investigator, Karen Elkind-Hirsch, Director of Research, Woman's
Other Study IDs: 05-013
Record Dates: First submitted 2008-05-28; First posted 2008-05-30 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-12

CONDITIONS: Gestational Diabetes Mellitus
Keywords: insulin sensitivity; insulin secretion; infant outcome
MeSH Terms: conditions — Diabetes, Gestational; Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples for insulin measurements
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1-NGT: normal glucose tolerance
- 2-GDM: Gestational Diabetes mellitus
- 3.GIGT: Gestational Impaired glucose tolerance

SUMMARY:
The project objective is to validate a new indirect estimate of insulin status in both pregnant African-American women and Caucasian women in southern Louisiana who are at risk for gestational diabetes mellitus. There are racial differences in carbohydrate metabolism that are potentially linked to complications during pregnancy and to increased risks of obesity and diabetes in later life. The investigators will explore the use of indexes of insulin status to identify the metabolic risk profile of pregnant women which may vary by race. Understanding whether there are differences which vary by race may influence clinical screening and treatment of pregnant women.

DETAILED DESCRIPTION:
The major goal of our proposed study is to validate a new approach to estimating insulin sensitivity and ß-cell function in African-American women compared to non-Hispanic white women in southern Louisiana who are at a high risk for gestational diabetes mellitus (GDM). We will determine whether the whole body insulin sensitivity index (WBISI) and insulinogenic index (IGI) [derived from an oral glucose tolerance test (OGTT)] can be used during 24-28 weeks of pregnancy to accurately estimate the degree of insulin resistance relative to ß-cell function in women with GDM in those with impaired glucose tolerance (IGT) as well as those who are glucose tolerant. Fasting values will also be assessed using the homeostasis model assessment (HOMA-IR and HOMA-%B) to evaluate insulin resistance and ß-cell function. We will explore the potential use of these measures to define the metabolic risk profile of these pregnant women and compare them with obstetric outcomes. We will determine if there are differences in risk that vary by race. Second, given the high likelihood that women who manifest GDM will develop type 2 diabetes mellitus (DM), identification of these patients by ethnic group or other independent determinants will permit intervention after delivery that might delay or prevent the onset of type 2 DM.

ELIGIBILITY:
Inclusion Criteria:

* 18-42 years of age
* at 20-30 weeks of gestation
* Caucasian or African-American and non-users of medications known to influence carbohydrate metabolism.

Exclusion Criteria:

* <18 years or >42 years of age
* non-Caucasian or non-African-American ethnicity
* use of drugs that could interfere with glucose or insulin metabolism; or health problems such as diabetes mellitus or liver, heart, lung and kidney diseases

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy, nondiabetic pregnant African-American and Caucasian women who have been scheduled for a standard 3-hour glucose tolerance test at 24-28 weeks in the Woman's Hospital Pathology laboratory.
Sampling Method: Non-Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2006-01; Primary Completion 2009-08 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Insulin action measures | 20-30 weeks of pregnancy

SECONDARY OUTCOMES:
infant gestational age | time of delivery

CONTACTS AND LOCATIONS:
Overall Officials: Karen E Elkind-Hirsch, Ph.D., Principal Investigator — Woman's Health Research Institute; Beverly Ogden, MD, Principal Investigator — Woman's Pathology Laboratory
Locations (1):
- Woman's Hospital Pathology Laboratory, Baton Rouge, Louisiana, United States

REFERENCES:
- [Background] Kirwan JP, Huston-Presley L, Kalhan SC, Catalano PM. Clinically useful estimates of insulin sensitivity during pregnancy: validation studies in women with normal glucose tolerance and gestational diabetes mellitus. Diabetes Care. 2001 Sep;24(9):1602-7. doi: 10.2337/diacare.24.9.1602. PMID 11522706